CLINICAL TRIAL: NCT05528965
Title: Parallel Versus Perpendicular Technique for Genicular Radiofrequency Ablation
Brief Title: Parallel Versus Perpendicular Technique for Genicular Radiofrequency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Halil Cihan Kose, Principal investigator, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 139/27
Record Dates: First submitted 2022-09-01; First posted 2022-09-06 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perpendicular Group (Experimental): Perpendicular genicular radiofrequency application
  Interventions: Procedure: Perpendicular Group
- Parallel Group (Active Comparator): Parallel genicular radiofrequency application
  Interventions: Procedure: Parallel Group

INTERVENTIONS:
Procedure: Perpendicular Group — Radiofrequency ablation was applied to the perpendicular group by placing the tip of electrode perpendicularly to contact the genicular nerves.
  Arms: Perpendicular Group
Procedure: Parallel Group — Radiofrequency ablation was applied to the parallel group by placing the electrode lay parallel to contact the genicular nerves.
  Arms: Parallel Group

SUMMARY:
Although there are different ways of performing genicular nerve radiofrequency on knee pain, to our knowledge, there is no stuies comparing the clinical outcomes of a parallel technique vs. a perpendicular technique. We aimed to compare the effectiveness of these both techniques.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Intra-articular injections in the knee during the 3 months prior to procedure
* Chronic pain syndrome
* Lumbar radicular pain
* Patients who are unwilling or mentally incapable to complete the study questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-05 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-09-15 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with a pain reduction of at least 50% compared to baseline expressed by the numerical rating scale (NRS) | 6 months after intervention.
  The proportion of patients with a pain reduction of at least 50% compared to baseline expressed by the numerical rating scale (NRS) (0-10).The lower the score, the least pain the patient experiences.

SECONDARY OUTCOMES:
The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 6 months after intervention.
  WOMAC is a 24-item scale under the headings of pain, stiffness and functional activity. Patients rate the amount of strain, pain felt, and joint stiffness during daily activities between 0 and 4 (0 is the best, 4 is the worst), and the total score is between 0 and 96.

CONTACTS AND LOCATIONS:
Locations (1):
- Health Science University Diskapi Yildirim Beyazıt Training and Research Hospital, Yenimahalle, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No